CLINICAL TRIAL: NCT04750915
Title: NIH-AARP Diet and Health Secondary Research Study Based on OH95CN025 Data
Status: Active, not recruiting | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10000195; 000195-C
Record Dates: First submitted 2021-02-10; First posted 2021-02-11 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04-10

CONDITIONS: Cancer; Mortality; Chronic Diseases
Keywords: Nutrition; Prospective Cohort; Lifestyle Factors; Cancer; Mortality; Natural History
MeSH Terms: conditions — Neoplasms; Chronic Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- AARP: Members of AARP, aged 50-71 years and who resided in one of six states or in two metropolitan areas in the United States

SUMMARY:
Background:

The NIH and the American Association of Retired Persons (AARP) conducted a Diet and Health Study. It studied the links between diet, cancer, and cause of death in a group of middle-aged people in the U.S. Researchers want to learn more about how diet and lifestyle can affect cancer and mortality.

Objective:

To clarify links between diet, lifestyle, cancer, death, and chronic diseases.

Eligibility:

AARP members ages 50 to 71 who took part in study #OH95CN025 and lived in California, Florida, Pennsylvania, New Jersey, North Carolina, Louisiana, Atlanta, or Detroit in 1995 1996.

Design:

This study will use existing data and samples. Participants will not be contacted.

Participants personal data, like name, date of birth, and address, will be used. This data will be kept private. Their data and samples will get a unique ID.

Data from other follow-up studies will be used.

Cancer outcome data will be obtained from the 8 sample areas. Many participants have moved to Arizona, Nevada, and Texas. Data will be obtained from those states as well.

Cause of death and date of death will be obtained from the National Death Index.

Cheek swab samples were gathered from 2004 to 2005. They will be used to study the oral microbiome.

The University of Washington (UW) will be added as a study site. UW will study air pollution.

The process of linking with the Virtual Pooled Registry Cancer Linkage System will be explored. It uses one system. Right now, 11 state systems are used to get and link data.

Paper records will be stored in locked file rooms. Electronic data will be stored on secure servers.

DETAILED DESCRIPTION:
Study Description

The purpose of this study is to analyze the data that have been collected as part of NIH-AARP study (OH95CN025), a historical cohort; in this study we seek to continue to conduct research, but no new study activities will be requested from the study participants.

Objective

To examine relationships between diet, lifestyle, and cancers by means of a prospective cohort design

To examine relationships between diet, lifestyle, and mortality by means of a prospective cohort design

To examine relationships between diet, lifestyle, and chronic diseases

Study Population

Data and samples from 566,398 members of the AARP (formally the American Association of Retired Persons), aged 50-71 years, and who resided in one of six states (California, Florida, Pennsylvania, New Jersey, North Carolina, and Louisiana) or in two metropolitan areas (Atlanta, Georgia and Detroit, Michigan) in 1995-1996

ELIGIBILITY:
* INCLUSION CRITERIA:
* AARP members
* aged 50 to 71 years
* resided in one of six states (California, Florida, Pennsylvania, New Jersey, North Carolina, and Louisiana) or in two metropolitan areas (Atlanta, Georgia and Detroit, Michigan) in 1995-1996

Ages: 50 Years to 71 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Members of the AARP (formally the American Association of Retired Persons), aged 50-71 years, and who resided in one of six states (California, Florida, Pennsylvania, New Jersey, North Carolina, and Louisiana) or in two metropolitan areas (Atlanta, Georgia and Detroit, Michigan) in 1995-1996.
Sampling Method: Non-Probability Sample
Enrollment: 566398 (Actual)
Dates: Start 2021-02-09 (Actual); Primary Completion 2050-12-31 (Estimated); Study Completion 2050-12-31 (Estimated)

PRIMARY OUTCOMES:
Incident Cancer | 12/31/2030
  All cancers
Chronic Diseases | 12/31/2030
  Chronic diseases
All cause and disease specific mortality (especially cancer) | 12/31/2030
  All cause and disease specific mortality

CONTACTS AND LOCATIONS:
Overall Officials: Rashmi Sinha, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States